CLINICAL TRIAL: NCT02176291
Title: Incomplete Response in Late-Life Depression: Getting to Remission With Buprenorphine
Acronym: IRLGREY-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jordan F. Karp (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Jordan F. Karp, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO13120236; R34MH101371 (NIH)
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Depression; Major Depressive Disorder
Keywords: Buprenorphine; Receptors, opioid; Receptors, opioid kappa and mu
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Buprenorphine; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buprenorphine (Experimental): Buprenorphine
  Interventions: Drug: Buprenorphine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Buprenorphine — low-dose buprenorphine (range 0.2 mg/day -- 2.0 mg/day)
  Other Names: suboxone; buprenex; temgesic; subutex
  Arms: Buprenorphine
Drug: Placebo — matched placebo
  Arms: Placebo

SUMMARY:
The purposes of this project are to examine the feasibility, safety, tolerability and clinical effect of low-dose buprenorphine as a novel treatment for late-life treatment-resistant depression and to develop preliminary data about mechanism of action.

DETAILED DESCRIPTION:
Up to one half of older patients with major depression develop Late-Life Treatment Resistant Depression (LL-TRD). Consequences of LL-TRD include suicide, worsened medical conditions, increased caregiver burden, and higher all-cause mortality. The development and testing of novel-mechanism pharmacotherapies is a public health priority embraced by National Institute of Mental Health (NIMH). Among the neuropeptidergic transmitters, opioids are known to modulate mood, and this system is often altered in patients with major depression. Targeting the opiate system in LL-TRD may positively modulate a system in which there is age-associated imbalance between circulating opiates and the density and binding affinity of mu and kappa opiate receptors. Buprenorphine (BPN) is an antagonist at the kappa opiate receptor and a partial agonist at the mu opiate receptor. Either, or both, of these pharmacodynamic actions may underlie its putative antidepressant effects. Our research group has open pilot data from 15 older adults with prospectively demonstrated treatment resistance to venlafaxine who were exposed to low-dose BPN, suggesting a clinically meaningful antidepressant effect. In addition, since BPN: 1) is available in sublingual formulation and 2) has a favorable safety and pharmacokinetic profile, it is an attractive candidate to re-purpose as a molecule for LL-TRD. Thus, the overarching aims of this project are to examine the feasibility, safety, tolerability and clinical effect of low-dose BPN as a novel treatment for LL-TRD and to develop preliminary data about mechanism of action (MOA).

The overarching aims are to examine the feasibility, safety, and tolerability of buprenorphine (BPN) as a novel treatment for late-life treatment resistant depression (LL-TRD). This also involves using translational tools of modern neurobiology (fMRI) to rapidly obtain proof-of-concept support for further clinical development. Formal dosing schedules in the use of buprenorphine have yet to be thoroughly established. This study hopes to determine optimal dosing strategies to improve acceptability.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= to 50 years.
2. Major depressive disorder (MDD), single or recurrent, as diagnosed by the Structured Clinical Interview for the DSM IV (SCID-IV).
3. Montgomery-Åsberg Depression Rating Scale (MADRS) >/= to 15.
4. Has or agrees to establish a clinical relationship with primary care physician (PCP).
5. Availability of an informant (e.g., emergency contact).

Exclusion Criteria:

1. Inability to provide informed consent.
2. Depressive symptoms not severe enough i.e.,Montgomery-Åsberg Depression Rating Scale ( MADRS) < 15 at the baseline assessments.
3. Dementia, as defined by The Modified Mini-Mental State (3MS) examination < 84 and clinical evidence of dementia (e.g., memory impairment, executive dysfunction, agnosia, apraxia, aphasia, with functional impairment).
4. Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms, as diagnosed by the Structured Clinical Interview for DSM (SCID).
5. Abuse of or dependence on alcohol or other substances within the past 3 months as determined by SCID, and confirmed by study physician interview.
6. Alcohol use amounting to 15 or more drinks per week or drinking 5 or more drinks on one occasion during any given week.
7. High risk for suicide (e.g., active suicidal ideation (SI) and/or current/recent intent or plan) AND unable to be managed safely in the clinical trial (e.g., unwilling to be hospitalized). Urgent psychiatric referral will be made in these cases.
8. Contraindication to venlafaxine extended release (XR) or BPN as determined by study physician including history of intolerance of either venlafaxine XR or BPN in the study target dosage range (venlafaxine XR at up to 300 mg/day; BPN at up to 2 mg/day).
9. Inability to communicate in English (i.e., interview cannot be conducted without an interpreter; subject largely unable to understand questions and cannot respond in English).
10. Non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).
11. Unstable medical illness, including delirium, uncontrolled diabetes mellitus, hypertension, or cerebrovascular or cardiovascular risk factors that are not under medical management. This will be determined based on information from the patient's personal physician and study physician's clinical judgment. Referral to the patient's personal physician or to a general practitioner will be made in these cases. Sodium and glucose levels done in the past 6 months are also reviewed before a subject begins study medication to determine if an illness is stable or uncontrolled. Individual lab parameters may deviate from normal without any associated pathophysiology or negative clinical affect; therefore we will follow the guide below before beginning starting any study medication.

    Sodium value of 135 but asymptomatic= consider to be normal and proceed without further testing.

    Sodium value of 134= repeat sodium. If value continues to be at 134 or higher and subject is asymptomatic, continue study participation but recheck sodium level after one week of exposure to study medication to confirm it has stayed stable.

    Sodium value of 133 or less= will evaluate subject's medication list to suggest possibly removing other medications which may be contributing to low sodium (in collaboration with their PCP), suggest fluid restriction and require repeat sodium that is normal range prior to commencing study.

    Glucose < 275 and asymptomatic= stable to proceed but will communicate value to PCP with participants permission.

    (see exclusion #17 for information on hepatic function lab parameters)
12. Subjects taking psychotropic medications that cannot be safely tapered and discontinued prior to study initiation. The following exceptions are allowed if they have been taken at a stable dose for at least 4 weeks prior to study entry and there is not a plan to change the dose during the next 28 weeks: benzodiazepines up to 2 mg/d lorazepam equivalent; other sedative-hypnotics (e.g., zolpidem, zaleplon, eszopiclone); gabapentin if prescribed for non-psychiatric indication (e.g., neuropathy).
13. History of opiate abuse or dependence.
14. Severe pain, defined as >/= 7 on 0-10 numeric rating scale for pain.
15. Concomitant use of strong or moderate CYP3A4 inhibitor (indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketonazole, nefazodone, saquinovir, telithromycin, aprepitant, erythromycin, fluconazole, grapefruit juice, verapamil, diltiazem)
16. Refusal to stop all opioids (to avoid precipitating opioid withdrawal).
17. Hepatic impairment- aspartate aminotransferase (AST) /alanine aminotransferase (ALT) > 1.5 times upper normal. If AST and ALT are within 1.5 times the upper limit, and subjects are asymptomatic, they will be considered medically stable to participate
18. Estimated Glomerular Filtration Rate (GFR) < 20 ml/min.
19. Inability/refusal to identify a person as an emergency contact.
20. Pregnancy
21. Contraindications to MRI

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-08; Primary Completion 2017-04 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan F. Karp, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Buprenorphine | Placebo
Started | 20 | 11
Completed | 15 | 11
Not Completed | 5 | 0
Not completed — Death | 1 | 0
Not completed — non compliance with protocol | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine | Placebo | Total
Number analyzed (Participants) | 20 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (9.7) | 65.6 (7.5) | 65.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 12 | 8 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 16 | 11 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 11 | 31

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Measure of depression severity, range of 0-60
  We calculated the mean change in depression severity for both groups using baseline MADRS and week 8 MADRS scores.
  Greater mean change represents better outcome.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Buprenorphine: Buprenorphine: low-dose buprenorphine (range 0.2 mg/day -- 1.2 mg/day)
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 15 | 11
units on a scale
  Change in MADRS | 3.47 (8.94) | 4.09 (8.06)
  Final MADRS score | 16.93 (8.68) | 14.64 (9.41)

2. Secondary Outcome: Brief Symptom Inventory--Anxiety Subscale (BSI)
Description: Measure of Anxiety Theoretical Range 0-2.4 with lower numbers indicating a better outcome.
  We calculated the mean change in anxiety for both groups using Phase 1 week 12 time point (baseline) and Phase 2 week 8 time point (final time point).
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine | Placebo
Number analyzed (Participants) | 18 | 11
units on a scale
  Change in BSI | 0.07 (1.39) | 0.06 (0.80)
  Final BSI Score | 0.74 (0.94) | 0.64 (0.48)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 1 year and six months.
Arm/Group | Buprenorphine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/11
Serious Adverse Events (participants affected / at risk) | 2/20 | 2/11
Other Adverse Events (participants affected / at risk) | 12/20 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buprenorphine (N=20) | Placebo (N=11)
death (Cardiac disorders) | 1 | 0 — death was determined to be due to cardiac disease unrelated to study participation.
severe abdominal pain (Gastrointestinal disorders) | 0 | 1
nausea and hypertension (General disorders) | 1 | 0 — These two condition were listed as the reasons for hospitalization
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — hospitalization for pneumonia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Buprenorphine (N=20) | Placebo (N=11)
Lightheadedness (General disorders) | 4/19 | 1
Insomnia (General disorders) | 3 | 2
Drowsiness (General disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 5 | 2
Dry Mouth (General disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Increased Blood Pressure (Cardiac disorders) | 2 | 2
Increased pulse (General disorders) | 1 | 1
urinary frequency (Renal and urinary disorders) | 2 | 0
Falls (General disorders) | 1 | 1
Increased Sleep (General disorders) | 0 | 1
Sweating (General disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Blurred vision (General disorders) | 0 | 1
Decreased Libido (General disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Coughing (General disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 1
Yawning (General disorders) | 1 | 0
Weight gain (General disorders) | 0 | 1
Myalgia (General disorders) | 1 | 0
Increased plasma glucose level (Endocrine disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT02176291/Prot_002.pdf
  • Statistical Analysis Plan (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT02176291/SAP_003.pdf